CLINICAL TRIAL: NCT01811511
Title: Efficacy and Safety of Chungkookjang on Improvement of Metabolic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Sun Park, Obesity Research Center of Chonbuk National University, Chonbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: ORC-MS-CKJA
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — chungkookjang

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chungkookjang (Experimental): Chungkookjang(35g/day)
  Interventions: Dietary Supplement: Chungkookjang; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): Placebo(35g/day)
  Interventions: Dietary Supplement: Chungkookjang; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Chungkookjang
  Other Names: Chungkookjang(35g/day)
Dietary Supplement: Placebo
  Other Names: Placebo(35g/day)

SUMMARY:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled crossover human trial to evaluate the efficacy and safety of chungkookjang on improvement of metabolic syndrome. The investigators measured decrement of body fat parameters, including Body Fat Mass, Percent Body Fat, Fat Free Mass, Weight and BMI(body mass index), and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-29 years old
* BMI(body mass index) ≥ 23 kg/m2 or WC(Waist Circumference) ≥ 90(men), WC(Waist Circumference) ≥ 85(women)
* Able to give informed consent

Exclusion Criteria:

* Allergic or hypersensitive to any of the ingredients in the test products
* The diagnosis of type 1 and type 2 diabetes or fasting glucose ≥ 126mg/dL
* Systolic pressure ≥ 160mmHg, diastolic pressure ≥ 100mmHg
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in Body Fat Mass | 12 weeks
  Body Fat Mass was measured in study visit 1(0 week) and visit 3(12 week).
Changes in Percent Body Fat | 12 weeks
  Percent Body Fat was measured in study visit 1(0 week) and visit 3(12 week).

SECONDARY OUTCOMES:
Change in Glucose | 12 weeks
  Glucose was measured in study visit 1(0 week) and visit 3(12 week).
Changes in Cholesterol | 12 weeks
  Cholesterol was measured in study visit 1(0 week) and visit 3(12 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Obesity Research Center of Chonbuk National University, Jeonju, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Byun MS, Yu OK, Cha YS, Park TS. Korean traditional Chungkookjang improves body composition, lipid profiles and atherogenic indices in overweight/obese subjects: a double-blind, randomized, crossover, placebo-controlled clinical trial. Eur J Clin Nutr. 2016 Oct;70(10):1116-1122. doi: 10.1038/ejcn.2016.77. Epub 2016 Jun 15. PMID 27302672
- [Derived] Back HI, Ha KC, Kim HM, Kim MG, Yu OK, Byun MS, Jeong DY, Jeong SY, Cha YS, Park TS. The influence of the Korean traditional Chungkookjang on variables of metabolic syndrome in overweight/obese subjects: study protocol. BMC Complement Altern Med. 2013 Oct 31;13:297. doi: 10.1186/1472-6882-13-297. PMID 24171779